CLINICAL TRIAL: NCT01104727
Title: Multi-Port vs. Single-port Cholecystectomy
Brief Title: Multi-Port Versus Single-port Cholecystectomy
Acronym: MUSIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: European Association for Endoscopic Surgery (Other)
Responsible Party: Principal Investigator, Alberto Arezzo, Assistant Professor of Surgery, European Association for Endoscopic Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAES-3
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Cholelithiasis
Keywords: SINGLE PORT SURGERY; LAPAROSCOPY, CHOLECYSTECTOMY
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multi port (Active Comparator): 4-Ports Cholecystectomy (4PC): a 12mmHg pneumoperitoeum is created either by a 10mm umbelical Hasson's port or by a Verress needle followed by a 10 mm umbelical port insertion; further one 10mm and two 5mm ports are placed according to the preferred technique. A straight or angulated laparoscope may be used. Laparoscopic graspers, monopolar hook, bipolar forceps, scissors and 10mm clips-applier are used. A plastic bag system might be used for gall bladder extraction if necessary. In both 10 and 12mm accesses, fascia is sutured with resorbable sutures. Skin is secured by either metallic agraffes or interrupted sutures.
  Interventions: Procedure: 4-Ports Cholecystectomy (4PC)
- Single port (Active Comparator): Single-Port Cholecystectomy (SPC): a 2.5cm long skin incision around the umbilicus is performed. The subcutaneous tissue is dissected, the muscular fascia exposed and incised along the middle line (linea alba) respecting the muscular tissue. Peritoneum is identified and incised. The Single-Port device is inserted and anchored.
  In order to retract the gallbladder a transcutaneous suture is placed in the right hypocondrium with a straight needle and a monofilament thread which are passed through the fundus and knotted outside the skin. The following steps reproduce the traditional laparoscopic cholecystectomy. Each centre will be left free to use dedicated instruments and which or traditional laparoscopic ones.
  Interventions: Procedure: Single-Port Cholecystectomy (SPC)

INTERVENTIONS:
Procedure: 4-Ports Cholecystectomy (4PC) — a 12mmHg pneumoperitoeum is created either by a 10mm umbelical Hasson's port or by a Verress needle followed by a 10 mm umbelical port insertion; further one 10mm and two 5mm ports are placed according to the preferred technique. A straight or angulated laparoscope may be used. Laparoscopic graspers, monopolar hook, bipolar forceps, scissors and 10mm clips-applier are used. A plastic bag system might be used for gall bladder extraction if necessary. In both 10 and 12mm accesses, fascia is sutured with resorbable sutures. Skin is secured by either metallic agraffes or interrupted sutures.
  Arms: Multi port
Procedure: Single-Port Cholecystectomy (SPC) — a 2.5cm long skin incision around the umbilicus is performed. The subcutaneous tissue is dissected, the muscular fascia exposed and incised along the middle line (linea alba) respecting the muscular tissue. Peritoneum is identified and incised. The Single-Port device is inserted and anchored.
  In order to retract the gallbladder a transcutaneous suture is placed in the right hypocondrium with a straight needle and a monofilament thread which are passed through the fundus and knotted outside the skin. The following steps reproduce the traditional laparoscopic cholecystectomy. Each centre will be left free to use dedicated instruments and which or traditional laparoscopic ones.
  Arms: Single port

SUMMARY:
The aim of this study is to compare results of the new surgical strategy to the traditional 4-ports technique for cholecystectomy in a randomized controlled trial (RCT). In particular we are going to investigate the procedures in terms of overall morbidity, while taking into considerations skin-incision's related morbidity, postoperative pain and cosmetic results which are the hypothetical benefits of the new approach. Other parameters are supposed to be unchanged, considering evidences from recent literature.

Surgical procedures:

4 ports cholecystectomy (4PC): a 12mmHg pneumoperitoeum is created either by a 10mm umbilical Hasson's port or by a Verress needle followed by a 10mm umbilical port insertion; further one 10mm and two 5mm ports are placed according to the preferred technique.

Single Port Access cholecystectomy (SPC): the single-port device is inserted through the umbilicus, by means of an adeguate incision, as the only access to the abdominal cavity. A trans-abdominal suture in right hypochondrium is placed through the gallbladder wall of the fundus to retract it.

Primary endpoint: overall morbidity rate (at 60 days from surgery)

Secondary endpoints:

1. skin-incision's related morbidity rate (at 60 days from surgery)
2. perioperative pain
3. cosmetic results
4. long-term morbidity (12 months)
5. intraoperative time
6. "conversion SPC to 4PC" rate
7. "conversion to laparotomy" rate
8. hospital stay

DETAILED DESCRIPTION:
Duration of the project Patients will be recruited for this study from September 2010 until September 2012 in all participating centers. All randomized patients will be followed up (after recovery) with outpatient clinic appointments 30 and 60 days from surgery. A long-term evaluation will be done 12 months after surgery. The last 3 months will be used for photographic analysis of cosmetic results, statistical analysis and reporting of data.

Hypothesis /Aims SPA technique is a feasible approach to the peritoneal cavity. While performing laparoscopic cholecystectomy the single umbilical access has an overall morbidity comparable to multiport laparoscopy (equivalence study) while it entails a reduced skin-incision's related morbidity rate, a reduced post-operative pain and allows a better cosmetic result. Other considered parameters (operative time, conversion rate and hospital stay) are supposed to be unchanged.

Background More recently Natural Orifice Translumenal Endoscopic Surgery (NOTES) has been highlighted to the attention of lay literature and media, after first clinical reports. Concept and feasibility had been tested in animal experiments since 20041, leading to the creation of new scientific societies and committees with the declared aim to regulate research activity, through sponsorships and registers, without reaching the goal completely. After less than three years, the race for the first cholecystectomy under NOTES conditions in a human being was having its course. Since then, many authors have reported various case collections, while many others presented consistent research activity in vitro or in vivo, but it looks evident that two different branches of research were being defined2 .

The first consists in what we would call Endoscopical Access Natural Orifice Surgery (EA-NOS) which includes all procedures truly performed through natural orifices, having the goal to design new platforms for surgery to be brought within the human body to recreate surgical conditions under safety. The evident difficulties to obtain such an environment with guaranteed ease of use, safety and efficacy, reduced to a mere research activity the interest in this field, with few clinical applications described consisting of hybrid procedures, i.e. procedures which were performed basically under laparoscopic conditions with the help of flexible instruments inserted through natural orifices. In fact, a recent large metanalysis of NOTES literature3 focusing on various surgical intra-abdominal procedures, all ascribable to EA-NOS, concluded that no human studies were found satisfactory for the inclusion criteria, for scarce disposable evidence, minor safety and efficacy compared to laparotomic and laparoscopic alternatives. The recommendation that human procedures should first pass through hybrid NOTES surgery, under strict guidelines, and in apposite controlled registers was later supported, as known, by the revision of NOSCAR "white paper" 4 . In fact, it is out of discussion that there is a need for a worldwide register, a standardization of the nomenclature, safety data to be used by ethical committees in order to authorize human trials, and implementation of the interface between medical societies, industry and regulatory offices. In this field, on behalf of the EURONOTES Foundation, we have promoted an european registry of NOTES procedures (www.euronotes.world.it) which preliminary results are now awaited.

The cooling of enthusiasm related to EA-NOS procedures has naturally forced surgeons to concentrate on techniques which could be more easily reproduced in clinical environments. This brought the interest towards what we would call Surgical Access Natural Orifice Surgery (SA-NOS)2 . In fact, an analysis of the literature would unveil that the vast majority of human studies can be ascribed to SA-NOS. A wider vision of what can be considered a SA-NOS approach, includes in this group not only transvaginal, thoroughly described in literature, but also trans-umbilical surgery. Although both approaches have the advantage of not being burdened by problems related to endoscopic defect's closure in terms of infection, safety, consistent technological research and time-consumption, there is no discussion that trans-umbilical techniques encountered more appreciation among surgeons. We have observed a rapid clinical diffusion driven by a technology development supported by all the different major surgical companies. Thus, it has to be said that single-port laparoscopic surgery is nothing new. It was 1992 when Marco Pelosi first described a laparoscopic appendectomy using a single umbilical puncture5 . Even multi-port single-incision trans-umbilical laparoscopic cholecystectomy was first described by Giuseppe Navarra already in 19977 . Despite this, interest towards single-port surgery grew-up only very recently. This might be on one side explained with the better establishment of laparoscopic techniques and skills over the years, but rises doubts about a possible industry driven interest.

There is no discussion that the technique has a number of drawbacks. The major one regards the concept of "triangulation" to which laparoscopic surgeons have grown accustomed in terms of both the instruments and scope, which is now lacking. Although this seems to be overshadowed by the increasing acceptability of in-line viewing, it has to be said that industries concentrate on developing and marketing a number of curved instrument with different characteristics with the aim of restoring standard triangulation as under laparoscopic environment. Nevertheless, personal experience gained by conducing a trial on a virtual reality simulator designed for the purpose, demonstrated that only very experienced surgeons performed surgical tasks with safety and effectiveness and requiring a short learning curve, while for all other surgeons technique acquisition was challenging7 .

Still a number of different concerns arise. The fundamental hypotheses that were at the base of single-port growing interest were that it could improve cosmesis, decrease post-operative pain and therefore probably allow an earlier return to work with in any case a better patient's satisfaction. None of these has been confirmed yet, if they will ever. It is also clear that those who advocate patients' preference as the main reason for proposing single-port techniques forget that patients' preference is deeply influenced by the assumption that these arguments in favor of single-port surgery are correct, despite there is no realistic certainty about it. Some of the major experts in the field of minimally invasive surgery and active researchers in the field of NOTES share the same skeptical opinion about a real benefit of single port techniques application. Dr Ratner for instance states in a recent interview that "...it is not clear to me whether single port laparoscopy would be beneficial compared to traditional laparoscopy"8 .

In any case we should never advocate for even slightly improved cosmetic value over safety, the principal concern. This has implications in both the intraoperative and the postoperative time. While it is recommended not to consider conversion to standard multi-trocars laparoscopy a failure, it might be that, as it happened at the beginning of the diffusion of laparoscopy, an increased number of complications will be observed. In fact, as often in similar circumstances, only a minority of efforts has been dedicated to training programs and very few simulators are available yet. Moreover, it has been advocated that a larger peri-umbilical incision and consequent fascial defect would imply a higher rate of incisional hernia. Although this is likely to happen, only time and data acquired will give us the answer.

For these reasons robust studies to show that there is indeed a difference without a significant compromise of safety should be awaited before a wide diffusion of these techniques. In the proposed study cholecystectomy is chosen as a target as it represent the typical and more diffuse indication for laparoscopy. Its morbidity rate related to skin incisions occurs in a range of 1 to 5%9,10.

REFERENCES Kalloo AN, Singh VK, Jagannath SB, Niiyama H, Hill SL, Vaughn CA, Magee CA, Kantsevoy SV (2004) Flexible transgastric peritoneoscopy: a novel approach to diagnostic and therapeutic interventions in the peritoneal cavity. Gastrointest Endosc 60(1):114-117 Vettoretto N, Arezzo A. Human natural orifice translumenal endoscopic surgery: on the way to two different philosophies? Surg Endosc. 2010 Feb;24(2):490-2.

Della Flora E, Wilson TG, Martin IJ, O'Rourke NA, Maddern GJ (2008) A review of natural orifice translumenal endoscopic surgery (NOTES) for intra-abdominal surgery: experimental models, techniques, and applicability to the clinical setting. Ann Surg 247(4):583-602 Hawes RH (2008) Transition from laboratory to clinical practice in NOTES: role of NOSCAR. Gastrointest Endosc Clin N Am 18(2):333-341 Pelosi MA, Pelosi MA 3rd. Laparoscopic appendectomy using a single umbilical puncture (minilaparoscopy). J Reprod Med. 1992 Jul;37(7):588-94.

Navarra G, Pozza E, Occhionorelli S, Carcoforo P, Donini I. One-wound laparoscopic cholecystectomy. Br J Surg. 1997 May;84(5):695 Rimonda R., Brown S., Tang B., Cuschieri A. Ergonomic performance with crossed and uncrossed instruments in single port laparoscopic surgery. Accepted for 12th SAGES (American Society of GastroEndoscopic Surgery) Congress, Washington DC (USA), April 2010; under review on Annals of Surgery.

Rattner D. Single port surgery and NOTES: competition or transition?. Epublication: WeBSurg.com, Nov 2007;7(11). URL: http://www.eats.fr/doi-vd02en2227rattner3e.htm Access-related complications - an analysis of 6023 consecutive laparoscopic hernia repairs. Minim Invasive Ther Allied Tecnol (2001) 1: 23-29 Hong T.H., You Y.K., Lee K.H. Transumbilical single-port laparoscopic cholecysectomy. Surg Endosc (2008) DOI 10.1007/s00464-008-0252-y

Study Design Design: multi-centric randomized controlled trial (RCT)

Primary endpoint: Overall morbidity rate defined as any diagnosed morbidity related to surgical technique within 60 days from surgery.

Primary outcome measure (for non-inferiority):

Morbidity, defined as the occurrence of any complication, directly or indirectly related to surgery. Complications will be classified according to Dindo [Dindo D., Demartines N., Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13)]

Complications will be subdivided into procedural (during treatment) and delayed complications (after ending the procedure), and further subdivided into major (requiring additional surgery) and minor (requiring endoscopic or medical intervention) complications.

During admission patients will be monitored for complications. The following standardized discharge criteria will be applied in all participating hospitals: normal intake of nutrition; normal mobility; absence of fever (<38°C); and stable hemoglobin level during 1 day (<1 mmol/L).

In case of same day discharge from the hospital patients will be called by telephone 1 day after the procedure whether adverse events have happened. Two weeks after the intervention, a research nurse will contact the patient by telephone again and ask for occurred complications.

The patient will undergo a direct check-up by means of a medical doctor at 30 and 60 days after surgery, to conclude evaluation.

Secondary endpoints:

Skin-incision related morbidity defined as bleeding, infection, necrosis, skin retraction, incisional hernia, suture dehiscence within 60 days from surgery.

Postoperative pain defined as a subjective evaluation of the same parameter using an horizontal visual analogical scale daily for the first week and weekly till 60 days after surgery. Patients will be administered Paracetamol IV 3 times a day for the first 24h, than on demand. Tramadol will be administered when Paracetamol will not be judged sufficient for pain control. On request, a single-dose of Ketorolac can be prescribed.

Cosmetic results defined as judgement of

* three independent surgeons: using a standardized methodology (patient on standing position against a black background), two digital photographs (JPG format, 800x600 pixels resolution, 16x106 colours, 24 bit) will be taken preoperatively (for comparison) and 60 days from surgery, one consisting of a close up of the umbilical area and a large view including just the full abdomen. A Likert scale will be used independently by the three surgeons to score the photographs from 1 to 5 (1= very poor, 2= poor, 3= satisfactory, 4= good, 5= very good) in all cases. The mean value will be considered objective evaluation of cosmetic outcome.
* the patient him/her self: the patient will be asked to score his/her subjective perception of cosmetic outcome using the same Likert scale 60 days from surgery.

A following comparison of the two different measures will give an interesting proportion of differences between subjective and objective perception.

Hospital stay: length (days) of hospital stay after surgery Intra-operative time: minutes between skin incision and end of skin closure Conversion "Single-Port (SPC) to Multi-Ports (4PC) Laparoscopy" rate: number of cases in which the surgeon preferred conversion from SPC to 4PC for safely of technical reasons Conversion "to Open Surgery" rate: number of cases in which the surgeon preferred conversion from SPC or 4PC to laparotomy for safely or technical reasons.

Long term morbidity defined as any diagnosed morbidity related to surgical technique within 1 year from surgery.

Patient recruitment: Consecutive eligible patients will be recruited at the outpatient clinic in the participating centres by the involved physician. All patients fulfilling the above-mentioned criteria will be informed about the study by the physician. After consent is given, central randomization will take place web-based and patients will be treated according to the study protocol. Patients unable or refusing to provide informed consent will be treated according to current clinical guidelines.

Randomization: patient data will be entered into a web-based database and a blind randomization (into two experimental groups: a. traditional 4-Ports Cholecystectomy (4PC) vs. b. Single-Port Cholecystectomy (SPC)) will be done by an unchangeable number-generating software.

Blinding: Blinding of patients and physicians during treatment is unfeasible, since the two treatment strategies are highly different and easily recognizable. Since a double-blinded method is not possible in surgical experiments, this system guarantees the highest scientific severity.

Study Population:

inclusion criteria: - age: 18-75

* BMI: <30 ASA: I-III absence of non-correctable coagulopathy (international normalized ratio >1,5, or platelet count <90 × 109/l).
* diagnosis: cholelithiasis (gallstones < 2 cm in diameter) gallbladder dyskinesia gallbladder polyps

exclusion criteria: - diagnosis: cholecystitis suspected presence of common duct stones suspected presence of biliary cancer Previous abdominal surgery Previous umbilical surgery

Intervention techniques:

4-Ports Cholecystectomy (4PC): a 12mmHg pneumoperitoeum is created either by a 10mm umbelical Hasson's port or by a Verress needle followed by a 10 mm umbelical port insertion; further one 10mm and two 5mm ports are placed according to the preferred technique. A straight or angulated laparoscope may be used. Laparoscopic graspers, monopolar hook, bipolar forceps, scissors and 10mm clips-applier are used. A plastic bag system might be used for gall bladder extraction if necessary. In both 10 and 12mm accesses, fascia is sutured with resorbable sutures. Skin is secured by either metallic agraffes or interrupted sutures.

Single-Port Cholecystectomy (SPC): a 2.5cm long skin incision around the umbilicus is performed. The subcutaneous tissue is dissected, the muscular fascia exposed and incised along the middle line (linea alba) respecting the muscular tissue. Peritoneum is identified and incised. The Single-Port device is inserted and anchored.

In order to retract the gallbladder a transcutaneous suture is placed in the right hypocondrium with a straight needle and a monofilament thread which are passed through the fundus and knotted outside the skin. The following steps reproduce the traditional laparoscopic cholecystectomy. Each centre will be left free to use dedicated instruments and which or traditional laparoscopic ones.

Complication/Intervention failure:

Conversion "single-port (SPC) to multi-ports (4PC) laparoscopy" is possible according to surgeon's decision, while performing the surgical procedure. Since the patients' recruitment is based on "intention to treat" the converted procedure will not be excluded from the study. Conversion rate will be considered as a relevant result of the experiment.

Similarly, conversion "to open surgery" both from 4PC and SPC is possible according to surgeon's decision, while performing the surgical procedure. Since the patients' recruitment is based on "intention to treat", the converted procedure won't be excluded from the study. Conversion rate will be considered as a relevant result of the experiment.

Sample size and Power calculation Assuming a baseline overall morbidity of 5% for both 4PC and SPC group (average morbidity based on specific literature) and considering a level of difference considered clinically significant of 0.05 (4.75 to 5.25%) for SPC to be non-inferior, with a β-error of 0.2 and α-error of 0.05, 300 patients are needed per randomization group.

600 patients in total allow to establish equivalence in terms of overall morbidity, with a statistical power of 80%. If the hypothesis is confirmed, secondary endopoints will eventually define benefits for the new surgical procedure in terms of reduced skin incision's related morbidity, lower postoperative pain and better cosmetic results.

The sample size calculation has been obtained by R-software (R Project for Statistical Computing, Lucent Technology, GNU General Public Licence) version 2.10.1, package epicalc, routine sample-size.

Data analysis Intra and post-operative results will be inserted in the web-based database at any time during the study by the recruiting surgeon. The photographic material will be up-loaded into the computed database as well; all patients' personal data will be considered strictly reserved in respect of privacy policy.

The Kolgoromow-test will be used to establish whether the results are parametric or not. According to data feature, T-Test/Chi-Square or Wilcoxon rank test will be used where appropriate. All analyses will be carried out primarily on an intention-to treat basis.

Impact on clinical practice and healthcare system SPA Surgery is an emergent frontier of surgical innovation and represents an alternative to multi-ports standard laparoscopy. The trans-umbilical technique allows to perform laparoscopy with the supposed benefit of reduced invasiveness. In recent literature a large number of studies have aimed to demonstrate feasibility and safety of the new method even if no randomized trial is still available for definitive conclusions. Once feasibility and safety will be shown we will have to investigate benefit for the patients. For these reasons we have chosen as primary endpoint overall morbidity while in order to demonstrate the supposed benefit (patient's reduced discomfort and better cosmetic outcome) and skin incision morbidity will be taken into consideration.

Since SPA surgical technique requires a consistent effort in terms of development of new technology and surgeon's adaptation, we consider this definition of primary relevance. As a matter of fact, a concrete introduction of SPA Surgery into daily practice is not possible without a concrete advantage for patients. Except one single trial comparing only postoperative pain (by Tsimoviannis et al. in G. Hatzikosta General Hospital, Ioannina Greece), at present there are no similar studies posted on USA and European trials databanks.

For these reasons, we believe the MUSIC trial should produce precious information with obvious recoils on clinical activity.

Track record of applicants including their experience in the field and any plot work carry out The present MUSIC project is the result of a collaboration between the members of EAES Technology Committee and the Board of the EAES. All applicants have big experience in the field of new technologies in laparoscopic surgery. In particular, many of them have taken part in development of new instruments and new techniques for trans-luminal endoscopic surgery (NOTES). Since SPA surgery is considered part of this new concept for a micro-invasive approach to the abdominal cavity, we consider their knowledge particularly useful in the coordination of the trial. Considering the high interest on SPA-surgery expressed in recent literature by the international surgical community, the Technology Committee has developed a specific interest in this new branch of surgical innovation.

Mario Morino, Alberto Arezzo. Video Surgery through Single Port Access: an overview. Revista Portuguesa de Cirurgia, in press Vettoretto N, Arezzo A. Human natural orifice translumenal endoscopic surgery: on the way to two different philosophies? Surg Endosc. 2010 Feb;24(2):490-2. Epub 2009 Jul 2.

Arezzo A, Kratt T, Schurr MO, Morino M. Laparoscopic-assisted transgastric cholecystectomy and secure endoscopic closure of the transgastric defect in a survival porcine model. Endoscopy. 2009 Sep;41(9):767-72. Epub 2009 Aug 14.

Arezzo A, Morino M. Endoscopic closure of gastric access in perspective NOTES: an update on techniques and technologies. Surg Endosc. 2010 Feb;24(2):298-303. Epub 2009 Jun 30.

Lirici MM, Arezzo A. Surgery without scars: the new frontier of minimally invasive surgery? Controversies, concerns and expectations in advanced operative endoscopy. Minim Invasive Ther Allied Technol. 2006;15(6):323-4.

Rimonda R., Brown S., Tang B., Cuschieri A. Ergonomic performance with crossed and uncrossed instruments in single port laparoscopic surgery. Accepted for 12th SAGES (American Society of GastroEndoscopic Surgery) Congress, Washington DC (USA), Aprile 2010; under review on Annals of Surgery.

Neugebauer EA, Becker M, Buess GF, Cuschieri A, Dauben HP, Fingerhut A, Fuchs KH, Habermalz B, Lantsberg L, Morino M, Reiter-Theil S, Soskuty G, Wayand W, Welsch T; On behalf of the EAES. EAES recommendations on methodology of innovation management in endoscopic surgery. Surg Endosc. 2010 Jan 7 Neugebauer EA, Morino M, Habermalz B. Surgical research or comic opera? Let's give answers! Surg Endosc. 2008 Jun;22(6):1411-2.

Meining A, Kähler G, von Delius S, Buess G, Schneider A, Hochberger J, Wilhelm D, Kübler H, Kranzfelder M, Bajbouj M, Fuchs KH, Gillen S, Feussner H.[Natural orifices transluminal endoscopic surgery (NOTES) in Germany: summary of the working group reports of the "D-NOTES meeting 2009"] Z Gastroenterol. 2009 Nov;47(11):1160-7 Fuchs KH, Breithaupt W. [Natural orifice transluminal endoscopic surgery in future obesity treatment] Chirurg. 2008 Sep;79(9):837-42.

Sylla P, Rattner DW, Delgado S, Lacy AM. NOTES transanal rectal cancer resection using transanal endoscopic microsurgery and laparoscopic assistance. Surg Endosc. 2010 Feb 26.

Lacy AM, Delgado S, Rojas OA, Ibarzabal A, Fernandez-Esparrach G, Taura P. Hybrid vaginal MA-NOS sleeve gastrectomy: technical note on the procedure in a patient. Surg Endosc. 2009 May;23(5):1130-7. MA-NOS radical sigmoidectomy: report of a transvaginal resection in the human. Surg Endosc. 2008 Jul;22(7):1717-23.

Project management structure

Once patients accept to be included in the MUSIC study, the randomization will be performed in one of the two groups:

1. Treatment A: 4 Ports Cholecystectomy (4PC)
2. Treatment B: Single-Port Access Cholecystectomy (SPC) Randomization will take place by connection to a dedicated web-site where initial data of the patient will be inserted and the group assignment will be displayed, sent by e-mail to the centre logged in and recruiting the patient, and stored in a dedicated database.

All the clinical informations related to the per-operative time and the follow-up as described in the appendix will be stored through the same website and collected in a database format. This will be accessible in an anonymous way, respecting the privacy of each patient, at any time. Basic statistical analysis as well as more advanced data analysis such as Wilcoxon tests and t-Student's test will be available online. Furthermore, the entire database can be downloaded at anytime in xls format for more advanced data analysis.

This will allow to complete an interim analysis and report to the Ethical committee at any time during the project. Proposed interval for analysis and reporting will be 3 months, if not suggested differently.

All applicants will be in charge of collection of data and analysis of results.

Dissemination plan Dissemination of research results, training and exploitation will be actively pursued. Results will be disseminated to the scientific community through specialized media, as selected magazines, conferences, fairs, websites and medical society, including clinicians considered final users and patients. Training activities will be carried out based on the dissemination activities, the target of the courses is expected essentially coming from the medical community.

The objective of the Dissemination Plan is to identify and organize the activities to be performed in order to promote the exploitation of the project's results and the widest dissemination of knowledge from the project.

MUSIC trial will establish an infrastructure for communications (and therefore dissemination) by building a robust framework in which dialogue and interaction can take place. This applies equally to internal and external communication. These will be used to disseminate information about and solicit input into the Single-Port-Access Surgery project work. Contact can be maintained and facilitated by electronic mailing lists, through Internal Lists within the EAES members, and External Lists including stakeholders using several existing lists to communicate to the wider community.

Moreover the MUSIC-working group develop a publications program which at minimum will comprise:

targeted informational literature designed to raise awareness about Single-Port-Access Surgery, and its activities instructional literature derived from experience across this trial, including methodological guidelines and strategic guides to good clinical practice.

The MUSIC-working group will develop effective mechanisms for dissemination material including the worldwide web, with a website which will include

* information about MUSIC study and its activities including contact details, background information, working papers, events (seminars, workshops, conferences) etc.
* instructional materials as discussed above n(the web in this respect acts as a principal means of publication):
* frequent news and updates to keep the community informed Finally printed publications will be submitted to the EAES Official Journal, Surgical Endoscopy.

The MUSIC-working group will be promoting dissemination, advocacy and other events. Conferences, workshops, seminars will be organized to:

raise awareness about activities, resources, results, etc.; act as training venues e.g. For disseminating instructional material as required by a particular stakeholding community or communities; act as for a for more public discussion of research, development, collections, standards or other strategic and substantive issues of interest to SPA Surgery and the wider community.

Long term sustainability of the work The program has the potential for long term sustainability according to its underlying concept.

Since Single-Port surgery is a traditional laparoscopy-like technique, the cost of procedure is expected to be similar. Other than different ports and instruments (already present on the market), SPC and 4PC require the same laparoscopic equipment, largely available in every operative room. From this point of view, the study doesn't imply any supplementary expense. The follow up of both procedures is identical. It will consist in outpatient clinical meetings and doesn't require expenses for new material and devices. Cost for complications and hospital stay is supposed to be unchanged between the two experimental groups.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-75
* BMI: <30
* ASA: I-III
* absence of non-correctable coagulopathy (international normalized ratio >1,5, or platelet count <90 × 109/l).
* diagnosis: cholelithiasis (gallstones < 2 cm in diameter) gallbladder dyskinesia

Exclusion Criteria:

* cholecystitis
* suspected presence of common duct stones
* suspected presence of biliary cancer
* Previous abdominal surgery
* Previous umbilical surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
overall morbidity rate (at 60 days from surgery) | 60 days
  Morbidity, defined as the occurrence of any complication, directly or indirectly related to surgery. Complications will be classified according to Dindo [Dindo D., Demartines N., Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13)]

SECONDARY OUTCOMES:
Skin-incision related morbidity | 60 days
  defined as bleeding, infection, necrosis, skin retraction, incisional hernia, suture dehiscence within 60 days from surgery.
Postoperative pain | 60 days
  defined as a subjective evaluation of the same parameter using an horizontal visual analogical scale daily for the first week and weekly till 60 days after surgery. Patients will be administered Paracetamol IV 3 times a day for the first 24h, than on demand. Tramadol will be administered when Paracetamol will not be judged sufficient for pain control. On request, a single-dose of Ketorolac can be prescribed.
Cosmetic results | 60 days
  * three independent surgeons: using a standardized methodology. A Likert scale will be used independently by the three surgeons to score the photographs from 1 to 5 (1= very poor, 2= poor, 3= satisfactory, 4= good, 5= very good) in all cases. The mean value will be considered objective evaluation of cosmetic outcome.
  * the patient him/her self: the patient will be asked to score his/her subjective perception of cosmetic outcome using the same Likert scale 60 days from surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Arezzo, MD, Study Director — European Association for Endoscopic Surgery
Locations (1):
- University of Turin, Torino, Italy

REFERENCES:
- [Derived] Arezzo A, Passera R, Bullano A, Mintz Y, Kedar A, Boni L, Cassinotti E, Rosati R, Fumagalli Romario U, Sorrentino M, Brizzolari M, Di Lorenzo N, Gaspari AL, Andreone D, De Stefani E, Navarra G, Lazzara S, Degiuli M, Shishin K, Khatkov I, Kazakov I, Schrittwieser R, Carus T, Corradi A, Sitzman G, Lacy A, Uranues S, Szold A, Morino M. Multi-port versus single-port cholecystectomy: results of a multi-centre, randomised controlled trial (MUSIC trial). Surg Endosc. 2017 Jul;31(7):2872-2880. doi: 10.1007/s00464-016-5298-7. Epub 2016 Oct 24. PMID 27778171
- [Derived] Steinemann DC, Raptis DA, Lurje G, Oberkofler CE, Wyss R, Zehnder A, Lesurtel M, Vonlanthen R, Clavien PA, Breitenstein S. Cosmesis and body image after single-port laparoscopic or conventional laparoscopic cholecystectomy: a multicenter double blinded randomised controlled trial (SPOCC-trial). BMC Surg. 2011 Sep 12;11:24. doi: 10.1186/1471-2482-11-24. PMID 21910897
- [Derived] Arezzo A, Morino M. Endoscopic surgery through single-port incision: time for a trial? Surg Endosc. 2011 Jun;25(6):1709-11. doi: 10.1007/s00464-011-1679-0. No abstract available. PMID 21553174